CLINICAL TRIAL: NCT02868060
Title: Evaluating the Pharmacokinetics and Pharmacodynamics of Romiplostim in Patients With Immune Thrombocytopenia (ITP)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin China Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 531-CN001
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Immune Thrombocytopenia (ITP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 mcg/kg AMG531 (Experimental): The administration of Romiplostim will be performed on Day 1 and 8
  Interventions: Drug: Romiplostim
- 3 mcg/kg AMG531 (Experimental): The administration of Romiplostim will be performed on Day 1 and 8
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim
  Other Names: AMG531

SUMMARY:
The objective of evaluating the pharmacokinetics and pharmacodynamics of romiplostim in patients with immune thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with immune thrombocytopenia (ITP) for at least 6 months prior to signing the informed consent form (ICF).
* Subject is ≥ 18 years old and ≤ 70 years old while signing the ICF.
* Patients who have no response or relapsed after splenectomy. Or patients who have not been splenectomised and have completed at least 1 prior treatment for ITP. Excluded having previously received recombinant human thrombopoietin (rHuTPO) or any other thrombopoietin receptor agonist.
* The mean of 3 scheduled platelet counts taken during the screening period must be: < 30 ×10^9/L, with none >35×10^9/L.

Exclusion Criteria:

* Any known history of bone marrow stem cell disorder. Any abnormal bone marrow findings other than typical of ITP.
* Any active malignancy. If prior history of cancer other than basal cell carcinoma or cervical carcinoma in situ, no treatment or active disease within 5 years prior to signing the ICF.
* Had received Eltrombopag, recombinant human thrombopoietin (rHuTPO) or other myeloproliferative leukemia (MPL) stimulation product.
* Received hematopoietic growth factors (e.g., granulocyte colony-stimulating factor, macrophage colony-stimulating factor, erythropoietin, interleukin-11) for any reason within 4 weeks prior to signing the ICF.
* Received any anti-malignancy agents (e.g., cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, interferon-alfa) for any reason within 8 weeks prior to signing the ICF.
* Received any monoclonal antibody drugs (e.g., rituximab) for any reason within 14 weeks prior to signing the ICF.
* Less than 4 weeks since end of any clinical trials about therapeutic drug or device for any indication prior to signing the ICF.
* Pregnant or breast feeding.
* In the opinions of the principal investigator or investigators, the patients are not suitable for participation in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-09; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
The incidence of all adverse events including evaluation of antidrug antibody status | Up to 43 days after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Chinese academy of medical science hematology hospital, Principal Investigator — Chinese academy of medical science hematology hospital
Locations (5):
- China (5):
  - Peking Union hospital, Beijing
  - West China hospital, Chengdu
  - Chinese academy of medical science hematology hospital, Tianjin
  - Wuxi People's Hospital, Wuxi
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Qi J, Zheng L, Hu B, Zhou H, He Q, Liu H, Kawai H, Yang R. Pharmacokinetics, Safety, and Pharmacodynamics of Romiplostim in Chinese Subjects With Immune Thrombocytopenia: A Phase I/II Trial. Clin Pharmacol Drug Dev. 2022 Mar;11(3):379-387. doi: 10.1002/cpdd.1059. Epub 2021 Dec 17. PMID 34921514